CLINICAL TRIAL: NCT04955743
Title: A Multicenter Phase 2 Trial to Evaluate Intracranial Response to Pembrolizumab and Lenvatinib in Patients With Brain Metastases From Melanoma or Renal Cell Carcinoma Who Are Anti-PD1/PD-L1 Experienced
Brief Title: Pembrolizumab and Lenvatinib in Patients With Brain Metastases From Melanoma or Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of activity in the drugs
Sponsor: Yale University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Harriet Kluger, Professor of Medicine, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000030391
Record Dates: First submitted 2021-06-28; First posted 2021-07-09 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Melanoma; Renal Cell Carcinoma; Brain Metastases; PD1/PD-L1 Experienced; Pembrolizumab; Lenvatinib; Metastatic Melanoma
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Brain Neoplasms | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: Melanoma (Experimental): Participants who are melanoma (PD-1/PD-L1-experienced)
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib
- Cohort 2: Renal Cell Carcinoma (Experimental): Participants who are Renal Cell Carcinoma (PD-1/PD-L1 experienced).
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg intravenous (IV) is administered every 3 weeks
Drug: Lenvatinib — 20 mg orally (PO) is administered daily

SUMMARY:
This is a phase 2, Simon's 2-stage designed study with 2 cohorts of anti-PD-1/PD-L1 experienced patients with untreated brain metastases: 1) melanoma and 2) renal cell carcinoma (RCC).

DETAILED DESCRIPTION:
This is a phase 2, Simon's 2-stage designed study with 2 cohorts of anti-PD-1/PD-L1 experienced patients with untreated brain metastases: 1) melanoma and 2) renal cell carcinoma (RCC). The primary endpoint of this study is to determine the best intracranial response of combined pembrolizumab and lenvatinib in patients with untreated brain metastases from melanoma or RCC who are anti-PD-1/PD-L1--experienced. Secondary endpoints include best overall objective response (combined intracranial and extracranial response), progression-free survival (PFS), overall survival (OS), duration of intracranial response, and rate of adverse events. Exploratory/correlative endpoints will include evaluation of pre-treatment tumor tissue (either intracranial or extracranial) for immunohistochemical markers (PDL-1, tumor infiltrating lymphocytes, and angiogenic factors) and genetic analysis of tumor mutations or mutational burden. Pre-treatment and on-treatment blood samples will be collected and evaluated for biomarkers of response by cytokine profiling and transcriptomic analysis.

Patients must have at least one evaluable asymptomatic intracranial lesion, no smaller than 5mm and no larger than 3 cm. Patients may have prior radiation to or surgical resection of a symptomatic brain metastasis as long as at least one untreated lesion or unequivocally growing lesion is present for response assessment. Pembrolizumab 200mg IV every 3 weeks will be administered in combination with lenvatinib 20 mg PO daily for up to 2 years.

Patients must have received at least 2 doses of an anti-PD-1/PD-L1 mAb at some point in their treatment course and must have unequivocal intracranial progression. Intracranial progression in patients who are anti-PD-1/PD-L1 experienced is defined as either development of a new brain lesion(s) or unequivocal progression in a previously irradiated or resected brain lesion(s) site. Patients can be deemed to have progression after discussion and group consensus of the case at tumor board. Secondary imaging assessments to confirm intracranial progression are not required.

Patients who are enrolled from sites outside of the Sponsor (Yale) must have patient eligibility approved by the Sponsor.

Archival tissue from extracranial and/or CNS metastases will be obtained, if available, for correlative studies. A baseline pre-treatment fresh biopsy will also be required from an accessible metastasis unless there is not an easily accessible site to biopsy or if a biopsy is determined to be unfeasible by the treating physician after discussion with the study PI. The tumor tissue will be studied retrospectively for PD-L1 expression, TIL characteristics, and other immune and angiogenic markers that may predict sensitivity to this drug combination.

First response assessment will be performed at 6 weeks and will include MRI of the brain and CT body scans (or other clinically indicated body imaging such as MRI or PET CT) to assess systemic disease. Brain metastasis response will be determined using modified RECIST (mRECIST) 1.1 criteria, and extracranial disease response will be determined using RECIST 1.1. Responses will be confirmed with repeat imaging done at 12 weeks. Subsequent imaging will be performed at 12-week intervals thereafter and include an MRI of the brain along with body imaging, which may include CT, MRI, or PET/CT, as clinically indicated. Patients will discontinue treatment for disease progression, unacceptable toxicity, patient withdrawal from the study, termination of study, or death. Patients may be treated beyond progression of intracranial metastases after consultation with the study PI, provided symptomatic lesions are treated with stereotactic radiosurgery (SRS) or surgery. Dose reduction of pembrolizumab for immune-related toxicities is not permitted. Dose-reduction of lenvatinib for related toxicities is permitted.

Number of Patients:

A total of up to 62 eligible patients will be enrolled (27 patients with melanoma with allowance for 3 additional patients if any are unevaluable and 29 patients with RCC with allowance for 3 additional patients if any are unevaluable). Either cohort can be stopped for futility according to Simon's two-stage design. The study will accrue for approximately 36 months and will be open for approximately 24 additional months as patients on study are followed.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of melanoma or RCC and untreated metastatic brain disease will be enrolled in this study.

   Male participants: A male participant must agree to use a contraception as detailed in the protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

   Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance per protocol during the treatment period and for at least 120 days after the last dose of study treatment.
2. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
3. Have histologic or cytologic confirmation from any body site of metastatic melanoma irrespective of BRAF mutation status or renal cell carcinoma irrespective of histologic subtype.
4. Patients who have had prior resection or biopsy of a CNS and/or extracranial metastasis will be required to provide a formalin-fixed, paraffin embedded (FFPE) specimen from tumor taken at the time of surgery, if available. Fresh biopsies of a metastatic lesion should be performed if clinically able.

   Note: Participants are not required to have new or repeat brain metastasis biopsies for enrollment on the trial.

   Note: For those who have never had CNS brain metastasis biopsies, tissue of an accessible extracranial lesion will be obtained pre-treatment, unless deemed not possible by the treating physician and upon discussion with PI. In this case, archival extracranial metastatic tissue will be suitable.
5. Have at least one brain metastasis that is at least 5 mm AND twice the MRI slice thickness, but less than or equal to 3 cm, which is asymptomatic, has not been previously radiated, and is not requiring immediate local therapy or steroids. Lesions situated in a previously irradiated area are considered allowed if measurable per the aforementioned criteria and if progression has been demonstrated. Patients with any lesion(s) >3 cm can be enrolled provided the following: (1) the lesion must receive local treatment prior to initiation of study drugs (either by stereotactic radiosurgery or resection), (2) the patient is not symptomatic from the lesion(s) once local therapy has been administered, and (3) at least one additional, non-treated lesion between 5 mm and 3 cm is still present.
6. Prior treatment for either the Melanoma or RCC cohorts may include: Patients must have received at least 2 doses of an anti-PD-1/PD-L1 drug at some point in their treatment course. Any number of prior treatments including PD-1/PD-L1 inhibitors are allowed. Anti-PD-1/PD-L1 does not have to be the most recent therapy. Patients with melanoma who developed brain metastasis within 6 months of the last dose of adjuvant anti-PD-1 can be enrolled.
7. Life expectancy of at least 3 months.
8. A history of radiotherapy for brain metastases is allowed up to 1 week before study treatment provided that neurologic sequelae are resolved, and that measurable untreated target lesion(s) remain.
9. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation.
10. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as a systolic BP ≤150 or a diastolic BP ≤90 mmHg at screening and on Cycle 1 Day 1.

    Note: Eligibility of a participant that is receiving ≥3 antihypertensive medications prior to study entry will require PI approval.
11. Have adequate organ function as defined in the protocol. Specimens must be collected within 10 days prior to the start of study treatment.

Exclusion Criteria:

1. Symptomatic melanoma or RCC brain metastases at the time of therapy initiation.
2. Active use of corticosteroids to control CNS symptoms, unless steroid requirement has been decreasing and currently on ≤10 mg of prednisone or its equivalent without CNS symptoms for 7 days or more.
3. Overt hemorrhage from CNS metastases.
4. Presence of leptomeningeal disease.
5. Unable to undergo MRI imaging (either due to such conditions as inability to lie flat for the scan duration, incompatible medical devices at risk for malfunction, and foreign metal objects that pose a safety risk for imaging).
6. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
7. Has received anti-cancer therapy including investigational agents within 14 days prior to allocation or less than 4 weeks from prior immunomodulating antibody (excluding anti-PD1/PD-L1).

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy, rash, and/or alopecia may be eligible.

   Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
8. Has received prior CNS radiotherapy within 1 week of start of study treatment. Participants must have recovered from all radiation-related toxicities and not require corticosteroids.
9. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
10. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

    Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
11. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
12. Has a known additional malignancy that is progressing or is requiring active treatment.
13. Has active autoimmune disease that has required systemic treatment in the past 3 months or a documented history of clinical severe autoimmune disease, or a syndrome that requires chronic systemic steroids or immunosuppressive agents. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency with prednisone < 10 mg or the equivalent, etc.) is not considered a form of systemic treatment. Subjects with thyroid disease or vitiligo will not be excluded from the study.
14. Has presence of gastrointestinal condition including malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
15. Has a pre-existing Grade ≥3 gastrointestinal or non-gastrointestinal fistula.
16. Serious non-healing or dehiscing wound.
17. Has radiographic evidence of major blood vessel invasion/infiltration. The degree of tumor invasion/infiltration of major blood vessels should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
18. Has clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study drug.
19. Has clinically significant cardiovascular disease within 6 months of the first dose of study intervention including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability.

    Note: Medically controlled arrhythmia is permitted.
20. Has prolongation of QTc interval (calculated using Fridericia's formula) to >480 msec.
21. New York Heart Association congestive heart failure of grade II or above, unstable angina, myocardial infarction within the past 6 months, or serious cardiac arrhythmia associated with significant cardiovascular impairment within the past 6 months.
22. Has urine protein ≥2 g/24-hour. Note: Participants with >1+ proteinuria on urine dipstick will undergo 24-hour urine collection for quantitative assessment of proteinuria.
23. Evidence of a bleeding diathesis, risk for severe hemorrhage, or clinically significant coagulopathy.
24. Uncontrolled hypertension (systolic BP >150 mmHg or diastolic BP >90 mmHg) in spite of an optimized regimen of antihypertensive medication.
25. Has a history of (non-infectious, non-radiation-induced) pneumonitis not responsive to steroids or has current pneumonitis. Patients will also be excluded if there are respiratory issues including active infection or require supplemental oxygen for activities of daily living.
26. Has an active infection requiring systemic therapy.
27. Has a known history of Human Immunodeficiency Virus (HIV).
28. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as a detectable qualitative HCV RNA level) infection.

    Note: No testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
29. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
30. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
31. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
32. Women of child-bearing potential who are unwilling to or unable to use an acceptable method of contraception to avoid pregnancy for the entire study and for at least 5 months after cessation of study drug or have a positive pregnancy test at screening or baseline, or who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Best brain metastasis response rate (BMRR) | up to 2 years from the start of treatment
  Best brain metastasis response rate (BMRR), defined as PR and CR per modified RECIST 1.1.

SECONDARY OUTCOMES:
Best overall objective response rate | up to 2 years from the start of treatment
  Best overall objective response rate, defined as Partial Response (PR) and Complete Response (CR) per RECIST 1.1.
Progression Free Survival (PFS) | up to 2 years from the start of treatment or to time of disease progression
  PFS, defined as the time from start of study drug administration to the date of the first documentation of disease progression or death from any cause, whichever occurs first.
Overall Survival (OS) | up to 2 years from the start of treatment or to time of death
  OS, defined as the time from start of study drug administration to date of death from any cause.
Duration of brain metastasis response | up to 2 years from the start of treatment
  Duration of brain metastasis response, defined as the time from response to the time of the first documentation of intracranial disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Kluger, MD, Principal Investigator — Professor of Medicine
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No